CLINICAL TRIAL: NCT01857544
Title: Phase 4 Study of Intravitreal Aflibercept Injection for Recalcitrant Central Retinal Vein Occlusion Associated Macular Edema Despite Prior Anti-Vascular Endothelial Growth Factor (VEGF) Therapy. (ARChiMEDES)
Brief Title: Study of Intravitreal Aflibercept Injection for Persistent CRVO-associated Macular Edema Despite Prior Anti-VEGF Therapy
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Tennessee Retina (Other)
Collaborators: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VGFT-OD-1313; VGFT-OD-1313 (Other: Regeneron Pharmaceuticals)
Record Dates: First submitted 2013-05-16; First posted 2013-05-20 (Estimated); Last update posted 2014-10-29 (Estimated); Status verified 2014-10

CONDITIONS: Retinal Vein Occlusion
Keywords: Retinal Vein Occlusion; Central Retinal Vein Occlusion; Macular Edema
MeSH Terms: conditions — Retinal Vein Occlusion; Macular Edema | interventions — aflibercept

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Aflibercept 2.0mg (Experimental): Single arm - Intravitreal Aflibercept 2.0mg, 0.05 milliliters, monthly for 6 months.
  Interventions: Drug: Aflibercept

INTERVENTIONS:
Drug: Aflibercept — Monthly 2.0mg Aflibercept Intravitreal Injection
  Other Names: VEGF-Trap; Eylea

SUMMARY:
The purpose of this study is determine the number of patients with complete resolution of macular edema secondary to central retinal vein occlusion following 6 monthly injections of Aflibercept.

DETAILED DESCRIPTION:
Twenty (20) consented participant who meet the inclusion criteria will be enrolled to be followed for 6 months. All subjects will receive monthly 2.0 mg intravitreal aflibercept injections.

ELIGIBILITY:
Inclusion Criteria:A patient must meet the following criteria to be eligible for inclusion in the study:

* Age >18 years
* Documented macular edema following central retinal vein occlusion
* Currently receiving treatment with intravitreal anti-VEGF therapy initiated at least 3 months months previously
* Documented intravitreal treatment with ranibizumab 0.5 mg (at least 3 doses, each one month apart) or bevacizumab 1.25 mg (at least 3 doses, each one month apart)
* Presence of persistent macular edema (defined as any of the following):

  * central foveal thickness (CFT) of > 300 microns by spectral-domain OCT
  * presence of any intraretinal or subretinal fluid
  * Receipt of intravitreal anti-VEGF injections more frequently than once per month
* Willingness and ability to comply with clinic visits and study-related procedures
* Ability to provide signed informed consent

Exclusion Criteria:

* Prior vitrectomy in the study eye
* Concurrent retinal vascular disease in the study eye that could compromise visual acuity or contribute to macular edema (e.g. diabetic retinopathy, age-related macular degeneration)
* Any concurrent intraocular condition in the study eye (e.g. diabetic retinopathy, advanced glaucoma) that, in the opinion of the investigator, could either

  * require medical or surgical intervention during the 6-month study period to prevent or treat visual loss; or,
  * if allowed to progress untreated, contribute to loss of at least 2 Snellen equivalent lines of best corrected visual acuity over the 6 month study period
* Active intraocular inflammation (grade trace or above) in the study eye, or history of idiopathic or autoimmune-associated uveitis in either eye
* Current vitreous hemorrhage in the study eye
* Active infectious conjunctivitis, keratitis, scleritis, or endophthalmitis in either eye
* Intraocular surgery (including cataract surgery) in the study eye within 60 days preceding baseline
* Systemic anti-VEGF treatment within the last 3 months prior to screening
* Prior intravitreal aflibercept injection in the study eye
* Macular laser photocoagulation within 4 months of screening
* Intravitreal or periocular corticosteroid within 4 months of screening
* Uncontrolled glaucoma in the study eye (defined as intraocular pressure ≥30 mmHg despite treatment with ocular antihypertensive medication)
* Allergy to fluorescein, povidone iodine (Betadine) or aflibercept
* Participation in a study of an investigational drug or device within 30 days prior to potential enrollment into the study
* Patients with cognitive dysfunction such as dementia, Alzheimer's disease or any other neuro-degenerative disorder.
* Pregnant or breast-feeding women
* Sexually active men* or women of childbearing potential** who are unwilling to practice adequate contraception during the study (adequate contraceptive measures include stable use of oral contraceptives or other prescription pharmaceutical contraceptives for 2 or more menstrual cycles prior to screening; intrauterine device; bilateral tubal ligation; vasectomy; condom plus contraceptive sponge, foam, or jelly, or diaphragm plus contraceptive sponge, foam, or jelly)

  * Contraception is not required for men with documented vasectomy. **Postmenopausal women must be amenorrheic for at least 12 months in order not to be considered of child bearing potential. Pregnancy testing and contraception are not required for women with documented hysterectomy or tubal ligation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2013-06; Primary Completion 2016-01 (Estimated); Study Completion 2016-03 (Estimated)

PRIMARY OUTCOMES:
Complete anatomic resolution of macular edema following central retinal vein occlusion (CRVO) as measured by Optical Coherence Tomography (OCT) | From baseline to Month 6

SECONDARY OUTCOMES:
Extent of reduction in macular thickness | Month 6
Extent of reduction in macular volume | Month 6
Mean change in best-corrected visual acuity (BCVA) | Month 6
Proportion of patients with gain or loss of 5, 10, and 15 letters in BCVA | Month 6
Number and severity of adverse events | 6 month-period

OTHER OUTCOMES:
Effect on macular leakage using fluorescein angiogram (FA) | Month 6
Effect on peripheral retinal non-perfusion | Month 6

CONTACTS AND LOCATIONS:
Overall Officials: Franco M Recchia, MD, Principal Investigator — Tennessee Retina, PC
Locations (1):
- Tennessee Retina, PC, Nashville, Tennessee, United States